CLINICAL TRIAL: NCT05836636
Title: Immune Monitoring of Prevalent Kidney Transplant Recipients Using Torque Teno Virus: A Single-Center, Prospective Cohort Study
Acronym: TTV-KTR-SGH
Status: Active, not recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/2170
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant Infection; Kidney Transplant Rejection; Kidney Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Torque teno virus DNA measurement — Torque teno virus DNA level will be obtained from all study subjects upon recruitment, when subjects are admitted and when subjects undergo kidney allograft biopsies.

SUMMARY:
Kidney transplant recipients (KTRs) suffer from immunosuppression-related adverse events (iRAEs), such as infections and malignancy from chronic immunosuppression exposure but are also at risk of graft loss from rejection with under-immunosuppression. Biomarkers that predict both iRAEs and rejection and allow individualisation of immunosuppression exposure are lacking. While plasma viral DNA levels of Torque Teno Virus (TTV), a widely prevalent, non-pathogenic virus, have been shown to predict both iRAE and rejection in incident KTRs within 1 year after transplant, its role for prevalent KTRs on stable immunosuppression is unclear.

The investigators hypothesise that plasma TTV levels can predict iRAEs and rejection in KTRs on stable immunosuppression and propose a pilot study to pursue three specific aims: (1) To determine the TTV levels and its relationship with clinical factors affecting the 'net state of immunosuppression' in prevalent KTRs. (2) To analyse the prognostic value of TTV levels for iRAEs and rejection in prevalent KTRs. (3) To compare the prognostic performance of TTV levels to commonly available biomarkers and composite prognostic scores.

The investigators seek pursue these aims by performing a single-centre, prospective, observational cohort study of 172 KTRs on stable immunosuppression for more than 3 months. TTV levels will be measured, using the TTV R-GENE® kit, upon recruitment and when kidney allograft biopsies are performed. Subjects will be monitored for iRAEs and rejection for at least 12 months.

The study will provide data on the distribution of TTV levels in a prevalent cohort of KTRs and analyse its relationship with clinical factors and important clinical outcomes. If the study indicates that TTV may be predictive of iRAEs and rejection, the investigators aim to conduct further studies including interventional studies using TTV levels to guide immunosuppression. Ultimately, the investigators aim to use TTV as a biomarker to optimise long-term immunosuppression exposure, reduce the risk of iRAEs without increase in rejection, and improve long-term outcomes for KTRs.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients on follow up at Singapore General Hospital (SGH)
* More than 21 years old
* On stable doses of immunosuppression for more than 3 months

Exclusion Criteria:

* Titration of immunosuppression (e.g. for rejection or infection) less than 3 months ago
* Active infection requiring treatment
* Less than 21 years old
* Unable to provide informed consent

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients (KTRs) on stable doses of immunosuppression for more than 3 months
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Severe infections defined as any infection requiring hospitalization | 1 year
  Any infection requiring hospitalization

SECONDARY OUTCOMES:
Opportunistic infections | 1 year
  intracellular bacteria, mycobacteria, Listeria monocytogenes, and Nocardia spp., herpesviruses (CMV, HSV, and VZV), polyomaviruses, yeasts (Candida and Cryptococcus), molds (invasive aspergillosis and mucormycosis), and parasites (Toxoplasma gondii, PJP, and Leishmania)
De novo malignancy | 1 year
  De novo malignancy
Calcineurin inhibitor nephrotoxicity (biopsy-proven) | 1 year
  Calcineurin inhibitor nephrotoxicity (biopsy-proven)
Rejection (biopsy-proven) | 1 year
  With and without borderline T cell-mediated rejection
Glomerulonephritis - de novo or recurrent (biopsy-proven) | 1 year
Graft function | 1 year
  serum creatinine, estimated glomerular filtration rate by the CKD-EPI equation and urine protein-to-creatinine ratio
Graft loss | 1 year
  Censored and non-censored for death
Mortality | 1 year
  All-cause and cause-specific - i.e., infection, malignancy, cardiovascular, others
Immunosuppression-related adverse event | 1 year
  Composite outcome of severe infections defined as any infection requiring hospitalization, opportunistic infections, de novo malignancy and calcineurin inhibitor nephrotoxicity
Immune-mediated adverse event | 1 year
  Composite outcome of rejection (biopsy-proven) and glomerulonephritis (biopsy-proven)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Ho QY, Lai CMD, Liew IT, Oon LLE, Lim KL, Chung SJ, Thangaraju S, Tien SC, Tan CS, Kee T. Immune monitoring of prevalent kidney transplant recipients using Torque Teno Virus: Protocol for a single-centre prospective cohort study. BMJ Open. 2023 Sep 19;13(9):e076122. doi: 10.1136/bmjopen-2023-076122. PMID 37730403